CLINICAL TRIAL: NCT07247396
Title: A Clinical Trial to Evaluate the Safety and Efficacy of CEA-Directed CAR-T Cell Immunotherapy in Patients With Advanced Colorectal Cancer and Peritoneal Metastases Following Cytoreductive Surgery
Brief Title: CEA CAR-T Therapy After Cytoreduction in Colorectal Cancer Patients With Peritoneal Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC101
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Peritoneal Metastases From Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal infusion of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-5x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells

INTERVENTIONS:
Biological: CEA-targeted CAR-T cells — Administration method: intraperitoneal infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This single-arm, open-label, dose-escalation trial aims to evaluate the safety and efficacy of CEA-targeted CAR-T cells and to obtain their pharmacokinetic profile in patients with advanced colorectal cancer and peritoneal metastases after cytoreductive surgery; the recommended dose will then be derived from these data.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation study to evaluate the safety, preliminary efficacy, and pharmacokinetics of CEA-targeted autologous CAR-T cells administered by intraperitoneal infusion in patients with advanced colorectal cancer and peritoneal metastases following cytoreductive surgery. Three dose levels will be tested: 1 × 10⁵, 3 × 10⁵, and 5 × 10⁵ CAR⁺ cells/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤75 years at the time of informed consent signing.
2. Pathologically confirmed colorectal cancer with peritoneal metastases.
3. Patients who have failed standard treatments (disease progression or intolerance, e.g., failure of oxaliplatin, irinotecan, fluorouracil, etc.) or have no effective treatment options.
4. Underwent cytoreductive surgery for peritoneal metastases from colorectal cancer, with cytoreduction completeness (CC) score of CC-0 to CC-2. Postoperative recovery is good, without severe postoperative complications. A baseline enhanced whole-abdominal CT scan (within 1 week before or after 1 month post-surgery) shows no distant metastases outside the peritoneum (e.g., liver, lung, bone, brain).
5. Tumor samples resected during cytoreductive surgery are confirmed CEA-positive by immunohistochemistry (distinct membranous staining, positive rate ≥10%).
6. Regardless of synchronous or metachronous peritoneal metastases, there are no metastatic sites outside the peritoneum, and the primary tumor has been resected.
7. Expected survival time of at least 3 months.
8. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
9. Unless otherwise specified, subjects must have adequate organ function as follows:

   1. Hematology: White blood cell (WBC) count ≥3.5×10⁹/L, neutrophil count ≥1.8×10⁹/L, lymphocyte count >0.5×10⁹/L, platelet count ≥80×10⁹/L, hemoglobin ≥90g/L.
   2. Cardiac function: Echocardiography shows left ventricular ejection fraction (LVEF) >50%, and electrocardiogram (ECG) shows no significant abnormalities.
   3. Renal function: Serum creatinine ≤2.0×ULN, blood urea nitrogen (BUN) ≤1.5×ULN.
   4. Liver function: ALT and AST ≤3.0×ULN; total bilirubin ≤2.0×ULN (≤3.0×ULN for Gilbert's syndrome).
   5. Oxygen saturation >92% without oxygen supplementation.
10. Women of childbearing potential have a negative pregnancy test within 7 days prior to enrollment, have no immediate plans for pregnancy, and agree to use contraceptive measures (or other fertility control methods) before and during the trial.
11. Male patients agree to use appropriate contraceptive methods.
12. Able to comply with the study protocol and follow-up procedures.

Exclusion Criteria:

1. Unwilling to sign the informed consent form.
2. Received or are currently receiving anti-tumor drug therapy within 2 weeks prior to enrollment, except for perioperative hyperthermic intraperitoneal chemotherapy.
3. Clinically confirmed active or uncontrolled bacterial, fungal, or viral infections.
4. Have other uncured malignant tumors, except for carcinoma in situ of the lung, carcinoma in situ of the cervix, or basal cell carcinoma of the skin.
5. Have a history of severe asthma, active autoimmune disease, immunodeficiency, or require long-term immunosuppressive drug therapy; exceptions include vitiligo, type 1 diabetes, autoimmune-related hypothyroidism requiring hormonal therapy, and psoriasis not requiring systemic treatment.
6. Have a history of mental illness.
7. Have uncontrolled comorbidities, including but not limited to symptomatic congestive heart failure, unstable angina, arrhythmia; severe coronary artery disease or cerebrovascular disease, or other diseases deemed ineligible by the investigator.
8. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with HBV DNA titer above the normal range; positive for hepatitis C virus (HCV) antibody with HCV RNA above the normal range; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis.
9. Known hypersensitivity to any component of the study product, or other potential hypersensitivity to immunotherapy as deemed by the investigator.
10. Pregnant or lactating women.
11. The investigator judges that the patient has other serious diseases that may affect follow-up and short-term survival.
12. Other situations deemed ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cell preparations in the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Safety and Tolerability] | From infusion through Month 3
  Incidence of adverse events during the study, evaluated per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) criteria
Obtained the recommended dose of CAR-T cells for the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Safety and Tolerability] | From infusion through Month 3
  Dose-limiting toxicity after CEA CAR-T cell infusion

SECONDARY OUTCOMES:
Peritoneal Progression-Free Survival(PPFS) of CEA CAR-T treatment in advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Effectiveness] | 2 years
  PPFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Progression-Free Survival(PFS) of CEA CAR-T treatment in advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Effectiveness] | 2 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CEA CAR-T treatment in advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Effectiveness] | 2 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)
Disease Recurrence/Metastasis Rate of CEA CAR-T treatment in advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Effectiveness] | 2 years
  The proportion of patients who experience disease recurrence or metastasis within a specified time period after CAR-T cell infusion.
To evaluate the toxicity related to CAR-T cell preparations in the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Safety] | From infusion through Month 3
  Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS): Graded according to ASTCT consensus criteria (Grade 1-5). The incidence of all grades and grade ≥3 toxicities, median onset time and duration, utilization rate of symptomatic treatments (e.g., corticosteroids), and temporal correlation between the occurrence of CRS and ICANS will be analyzed. On-target/off-tumor toxicity involving CEA-expressing organs: The incidence of gastrointestinal toxicity (e.g., oral mucositis, diarrhea, colitis) and pulmonary toxicity (e.g., immune-related pneumonia) will be evaluated.
To evaluate the long-term biosafety of CAR-T cell preparations in the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Pharmacokinetics] | From infusion through Month 3
  To determine the time to maximum observed concentration (Tmax) of circulating CAR-T cells.
To evaluate the long-term biosafety of CAR-T cell preparations in the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Pharmacokinetics] | From infusion through Month 3
  To estimate the area under the concentration-time curve from time 0 to 28 days (AUC₀-₂₈d) and from time 0 to 90 days (AUC₀-₉₀d) for circulating CAR-T cells.
To evaluate the long-term biosafety of CAR-T cell preparations in the treatment of advanced colorectal cancer with peritoneal metastases following cytoreductive surgery [Safety] | 2 years
  Immunogenicity: Incidence of anti-CAR antibodies will be assessed. Delayed toxicity: Occurrence of events such as secondary malignancies will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lifeng Sun, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Ying Yuan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No